CLINICAL TRIAL: NCT03698539
Title: The Interaction Between Stuttering and Gestures and Their Influence on the Intelligibility of Individuals With Down Syndrome
Brief Title: How Stuttering and Gestures Influence the Intelligibility of Individuals With Down Syndrome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Marguerite-Marie Delacroix (Unknown); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s62049
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Stuttering; Down Syndrome; Intelligibility, Speech; Gestures
Keywords: Stuttering; Down syndrome; Gestures; Intelligibility
MeSH Terms: conditions — Stuttering; Down Syndrome; Speech Intelligibility; Gestures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Down syndrome who stutter: This group consists of individuals with Down syndrome who stutter. They have a mild or moderate intellectual disability and are able to understand and produce a three word sentence.
  Spontaneous hand gestures and stutter frequency are investigated in this group.
  Interventions: Behavioral: hand gestures
- Down syndrome who do not stutter: This group consists of individuals with Down syndrome who do not stutter. They have a mild or moderate intellectual disability and are able to understand and produce a three word sentence.
  Spontaneous hand gestures are investigated in this group
  Interventions: Behavioral: hand gestures
- Typically developing children who stutter: This group consists of typically developing children who stutter. They function as a control group to the individuals with Down syndrome.
  Interventions: Behavioral: hand gestures
- Typically developing children who do not stutter: This group consists of typically developing children who do not stutter. They function as a control group to the individuals with Down syndrome.
  Interventions: Behavioral: hand gestures

INTERVENTIONS:
Behavioral: hand gestures — We observe the use of spontaneous hand gestures in all the groups.

SUMMARY:
This study wants to determine the relationship between spontaneous hand gestures, stuttering and intelligibility in individuals with Down syndrome. One third of these individuals has fluency problems, such as stuttering. Gesture use appears to be a strength in individuals with Down syndrome. While they are able to compensate for their language problems, it is not clear if they also use gestures to compensate for their speech problems. Therefore, this study will observe the impact of their gesture use on the stuttering frequency/severity and on the intelligibility of children with Down syndrome.

This study has three research questions. The first question is: Is there a difference in gesture use between individuals with Down syndrome who stutter and individuals with Down syndrome who do not stutter? The hypothesis is that the children who stutter will make more gestures to compensate for the fluency problems. The kind of spontaneous hand gestures will also be considered. These results will be compared to those of typical developing individuals.

The second research question is: Are stuttering events that are accompanied by a gesture more intelligible than stuttering moments that are not accompanied by a gesture? Research showed that the use of signs has an positive impact on the speech intelligibility of individuals with Down syndrome. Here it is investigated if this is also true for spontaneous hand gestures. In case of better speech intelligibility it is investigated if the gain in intelligibility is caused by how recognizable the gesture is or by the effect of the gestures on speech itself. The effect of different types on the speech intelligibility of the stuttering events will also be investigated. Typically developing individuals who stutter will function as control group.

The third research question is: 'Does gestural priming have an influence on the fluency of children with Down syndrome? Gestural priming is a secondary speech signal that gives feedback to the first speech signal by simultaneously mimicking the first speech signal. In this research a hand puppet will imitate the mouth movements of the participants. Next to that, the speech will be simultaneously be accompanied by beat gestures, meaningless up and downward movements. The hypothesis is that due to mirror neurons, the participants will become more fluent. Mirror neurons are neurons in the brain that can produce a neural basis for fluency by the perception of the second speech signal.

DETAILED DESCRIPTION:
The parents of the individuals with Down syndrome are given a questionnaire to see if their child can participate in the study. A receptive language test is administered to the individuals with Down syndrome to get an indication of their developmental age. An stuttering discrimination test and a stuttering awareness test were also developed for this study, to see if individuals with Down syndrome are able to hear the difference between stuttered and fluent speech and to see if they are aware of their stuttering. Awareness of stuttering might impact their gesture use.

For the first research question, the relationship between gestures on the stuttering frequency/severity is investigated. To collect this information, video's of spontaneous speech will be analyzed. All the participants are filmed by their parents or caregivers. During the spontaneous speech, the individuals talk about anything they want. Multiple video's with different subjects are filmed per participant since stuttering is very variable. For example, if a child is more excited by one topic than by another, it could increase the stuttering frequency. The same procedure is administered to typically developing individuals. The transcription program CLAN is used to transcribed the videos and to code the stuttering events and the gestures. After this, statistical analysis is used to see if individuals with Down syndrome who stutter differ in their gesture use from the individuals who do not stutter. Next to that, the results of the Down syndrome group will be compared to the typically developing group.

For the second research question, the videos of the individuals are used to investigate the effect of gestures on the intelligibility of stuttering events. There are two conditions: (1) Videos of stuttering events with and without a gesture and (2) audio recordings of stuttering events with and without a gesture (4).The audio recordings are identical to the information in the video recordings.

Typically developing adults who are naïeve to the research question are asked to watch or listen the video/audio recordings of the individuals with Down syndrome. For each recording they are asked to transcribe what they thought the individuals with Down syndrome had said and on a 7-point Likert scale they had to indicate how intelligible they found the speech. The intelligibility results are compared between gesture and no gesture and between audio and video.

The same protocol will be done with video/audio recordings of typically developing individuals who stutter and their results will be compared to those of the participants with Down syndrome.

For the third research question, only the group of children who stutter is retained. There are three experimental conditions and one control condition based on the procedure of Snyder, Waddell & Blachet (2016). In the control condition, the investigator shows three pictograms on a laptop that form a sentence, for example, the cat eats cake. The participants have to produce this sentence. There is a training session to make sure the participant understands to goal of the pictograms and can produce the sentences. The actual test condition contains 7 sentences. In the control condition no gestures or priming is used. The experimental conditions are the same, but priming is induced. In the first experimental condition, the participant gets a hand puppet that must make the same mouth movements as she does, but the puppet needs to start moving before the participant starts talking. In the second experimental condition, the participant does the same thing with the hand puppet, but she has to hold it behind a screen, so she cannot see it herself. In the third condition, it is the investigator who simultaneously mimics the participant with the hand puppet. Each participant does all the conditions, but in a different order, so there is control for a saturation effect. Each experimental condition is preceded by a training session where different forms of prompting are used to teach to participants how to work with the hand puppet.

Additionally, since it is unnatural to walk around with a hand puppet, the same experiment is executed but with the use of beat gestures. These are rhythmical gestures that control the parsing of the speech stream. The children produce the sentences again but this time they make simple up and downward beat gestures during their speech or watch the experimenter make these gestures while they speak. The second experimental condition is eliminated in this case, since beat gestures are often made with two hands.

All the conditions are videotaped and transcribed in CLAN. The stuttering frequency is measured for all the conditions and compared between them. If the beat gestures have a fluency inducing effect, than this might be an indication to develop a new stuttering therapy based on spontaneous hand gestures.

ELIGIBILITY:
Inclusion Criteria for the participants with Down syndrome

* Stuttering (group 1)
* No stuttering (group 2)
* Able to understand and produce a three-word sentence
* Mild to moderate mental disability

Exclusion Criteria:

* Severe mental disability
* No understanding and/or production of a three-word sentence
* Uncorrected visual or auditory impairment

Inclusion Criteria for the typically developing participants

* Stuttering (group 1)
* No stuttering (group 2)
* Able to understand and produce a three-word sentence

Exclusion Criteria:

* No understanding and/or production of a three-word sentence
* Uncorrected visual or auditory impairment
* Other language/speech problems

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The groups will be assembled from individuals with Down syndrome and typically developing children who do and do not stutter who live in Flanders. They will be recruited via regular and special education primary schools, via speech language pathologists, via revalidation centra and via the Down syndrome association Flanders.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Gesture frequency | This frequency is measured in the spontaneous telling task and in the gestural priming experiment over a period of 4 - 6 months.
  This frequency is calculated by adding up all the gestures used by the participant and dividing it by the total of words the participant said. Tis total is multiplied by 100 to get a percentage. For example, if a participant used 10 spontaneous hand gestures in a speech sample of 50 words, he has a spontaneous hand gesture frequency of 20%. The speech samples are defined by the length of the videos. Every outing of the participant is included in the sample.
Stuttering frequency | This frequency is measured for the first, and third research question, once per participant who stutters over a period of 4-6 months.
  This frequency is calculated for the children with Down syndrome who stutter. The total number of stuttering moments is divided by the total number of words in the speech sample. This number is multiplied by 100 to get the stutter frequency. For example, if a participant had 9 stuttering moments in a speech sample of 90 words, he would have a stutter frequency of 10%. Stuttering moments are defined by repetitions of short words, interjections, syllables or sounds, the prolongation of sounds and blockages. The stutter frequency is calculated in all the studies. The length of the videos defines the speech samples. Every outing of the participant is included in the sample.
Subjective Intelligibility | This frequency is measured for the second research question, over a period of two months.
  The intelligibility of the individuals who stutter is measured with a 7-point Likert scale with 1 = completely unintelligible to 7 = completely intelligible
Objective Intelligibility | This frequency is measured for the second research question, over a period of two months.
  The intelligibility of the individuals who stutter is measured by comparing what the listeners transcribed to the true transcription.

SECONDARY OUTCOMES:
Stuttering discrimination | This is measured once before the start of the first research question.
  The ability to discriminate between stuttered and fluent speech is measured by a new test developed by the researcher.
Stuttering awareness | This is measured once before the start of the first research question.
  Stuttering awareness is measures by a new test developed by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Zink, Professor, Principal Investigator — Experimental Oto-Rhino-Laryngology, Dept. Neursciences, KU Leuven; Bea Maes, Professor, Principal Investigator — Parenting and Special Education, Faculty of Psychology and Educational Sciences, KU Leuven; Ellen Rombouts, Professor, Principal Investigator — Experimental Oto-Rino-Laryngology, Department Neurosciences, KU Leuven; Babette Maessen, Master, Principal Investigator — Experimental Oto-Rino-Laryngology, Department Neurosciences, KU Leuven
Locations (1):
- Experimental Oto-Rhino-Laryngology, Departement Neurowetenschappen, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenwald CA, Leonard LB. Communicative and sensorimotor development of Down's syndrome children. Am J Ment Defic. 1979 Nov;84(3):296-303. PMID 160755
- [Background] Smith L, von Tetzchner S. Communicative, sensorimotor, and language skills of young children with Down syndrome. Am J Ment Defic. 1986 Jul;91(1):57-66. PMID 2943160
- [Background] Bray M, Is stuttering therapy useful for adolescents and adults with Down syndrome who are dysfluent. Procedia. 2015; 193:51-61.
- [Background] Kent RD, Vorperian HK. Speech impairment in Down syndrome: a review. J Speech Lang Hear Res. 2013 Feb;56(1):178-210. doi: 10.1044/1092-4388(2012/12-0148). Epub 2012 Dec 28. PMID 23275397
- [Background] Terminology pertaining to fluency and fluency disorders: guidelines. ASHA Special Interest Division 4: Fluency and Fluency Disorders. ASHA Suppl. 1999 Mar-Apr;41(2 Suppl 19):29-36. No abstract available. PMID 10188303
- [Background] Bijlsma EK, Oosterwijk JC, Leschot NJ, Geraerdts, JPM, Prok JC, editors. Leerboek medische genetica [Textbook medical genetics]. Maarssen: Elsevier gezondheidszorg; c2005. 430 p. (Cassiman JJ, Engelen JJM, editors. Chromosomale overerving [Chromosomal inheritance]; vol.6).Dutch
- [Background] Chapman RS (1997). Language development in children and adolescents with Down syndrome. Ment Retard Develop Dis Res Rev. 1997; 3: 307-312.
- [Background] Fletcher P, Macwhinney B, editors. The handbook of child language. Oxford,UK:Blackwell; c1995. 800 p. (Chapman RS, editor. Language development in children and adolescents with Down syndrome; vol. 3).
- [Background] Eggers K, Van Eerdenbrugh S. Speech disfluencies in children with Down Syndrome. J Commun Disord. 2018 Jan-Feb;71:72-84. doi: 10.1016/j.jcomdis.2017.11.001. Epub 2017 Nov 8. PMID 29129311
- [Background] Góral-Półrola J, Zielińska J, Jastrzebowska, G, Tarkowski, Z. Cluttering: Specific communication disorder. Acta neuropsych. 2015; 14(1): 1-15.
- [Background] Guitar B. Stuttering. An integrated approach to its nature and treatment.3re ed. Baltimore: Lippincott, Williams & Wilkins; 2006. 376 p.
- [Background] Hammond G, editor. Cerebral control of speech and limb movements. Amsterdam: North-Holland; c1990. 708 p. (Flanagan R, Feldman, A, Ostry. Control of human jaw and multi-joint arm movements; vol.1).
- [Background] Loncke F, Nijs M, Smet L. SMOG: Spreken Met Ondersteuning van Gebaren [SMOG: Speaking With Support of Signs].4th ed. Antwerpen: Garant; 2012. 180 p. Dutch
- [Background] Preus, A. Treatment of mentally retarded stutterers. J Fluency Dis. 1990; 15(4):223-233.
- [Background] Chapman RS. Language learning in Down syndrome: the speech and language profile compared to adolescents with cognitive impairment of unknown origin. Downs Syndr Res Pract. 2006 Jul;10(2):61-6. doi: 10.3104/reports.306. PMID 16869363
- [Background] Galeote M, Sebastian E, Checa E, Rey R, Soto P. The development of vocabulary in Spanish children with Down syndrome: comprehension, production, and gestures. J Intellect Dev Disabil. 2011 Sep;36(3):184-96. doi: 10.3109/13668250.2011.599317. PMID 21843033
- [Background] Roberts JE, Price J, Malkin C. Language and communication development in Down syndrome. Ment Retard Dev Disabil Res Rev. 2007;13(1):26-35. doi: 10.1002/mrdd.20136. PMID 17326116
- [Background] Pruess JB, Vadasy PF, Fewell RR. Language development in children with Down syndrome. Educ Train Ment Retard. 1987; 22(1): 44-55.
- [Background] St. Louis KO, Myers, FL. Clinical management of cluttering. Lang Speech Hear Serv Schools. 1995; 26(2): 187-195.
- [Background] Mayberry RI, Jaques J, DeDe G. What stuttering reveals about the development of the gesture-speech relationship. New Dir Child Dev. 1998 Spring;(79):77-87. doi: 10.1002/cd.23219987906. No abstract available. PMID 9507705
- [Background] Snyder GJ, Waddell DE, Blanchet P. Mirror neurons as a model for the science and treatment of stuttering. Neuroreport. 2016 Jan 6;27(1):56-60. doi: 10.1097/WNR.0000000000000500. PMID 26565808
- [Background] Saltuklaroglu T, Kalinowski J. The inhibition of stuttering via the perceptions and production of syllable repetitions. Int J Neurosci. 2011 Jan;121(1):44-9. doi: 10.3109/00207454.2011.536361. PMID 21171820
- [Background] Kalinowski J, Stuart A, Rastatter MP, Snyder G, Dayalu V. Inducement of fluent speech in persons who stutter via visual choral speech. Neurosci Lett. 2000 Mar 10;281(2-3):198-200. doi: 10.1016/s0304-3940(00)00850-8. PMID 10704777
- [Background] Willems RM, Hagoort P. Neural evidence for the interplay between language, gesture, and action: a review. Brain Lang. 2007 Jun;101(3):278-89. doi: 10.1016/j.bandl.2007.03.004. Epub 2007 Apr 9. PMID 17416411
- [Background] Schaerlaekens A. [Assessing and measuring language development in the child. The Reynell Scales in a Dutch language area]. Folia Phoniatr Logop. 1995;47(6):303-9. doi: 10.1159/000266367. German. PMID 8868934
- [Background] Velthuijs M. Een taart voor kleine beer [A pie for little bear]. Rijswijk: De Vier Windstreken;1995. 27 p. Dutch
- [Background] Meuris K, Maes B, Zink I. Evaluation of language and communication skills in adult key word signing users with intellectual disability: advantages of a narrative task. Res Dev Disabil. 2014 Oct;35(10):2585-601. doi: 10.1016/j.ridd.2014.06.020. Epub 2014 Jul 10. PMID 25016435
- [Background] Arenas, R. M. Conceptualizing and investigating the contextual variability of stuttering: The speech and monitoring interaction (SAMI) framework. Speech, Lang. Hear. 20, 15-28 (2017).
- [Background] Clibbens, J. & Powell, G. Actions speak louder than words: signing and speech intelligibility in adults with Down syndrome. Down Syndr. Res. Pract. 2, 127-129 (2007).
- [Background] Garcia JM, Cannito MP. Influence of verbal and nonverbal contexts on the sentence intelligibility of a speaker with dysarthria. J Speech Hear Res. 1996 Aug;39(4):750-60. doi: 10.1044/jshr.3904.750. PMID 8844555